CLINICAL TRIAL: NCT00998166
Title: A Phase 2 Study of Cisplatin + Pemetrexed + Avastin as First-Line Therapy in Patients With Advanced Non-Squamous, Non-Small Cell Lung Carcinoma
Brief Title: A Study of Cisplatin + Pemetrexed + Avastin as First-Line Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAB9652
Record Dates: First submitted 2009-10-14; First posted 2009-10-20 (Estimated); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pemetrexed, Cisplatin, Bevacizumab (Experimental): Chemotherapy infusion on Day 1 of a 3-week cycle
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Pemetrexed — 1. Pre-hydration for 1-1/2 hours at 250 ml/hour
  2. Pemetrexed 500 mg/m2 IV over 10 minutes
  3. Return to hydration for 30 minutes at 250 ml/hour
  Other Names: Alimta
Drug: Cisplatin — 4. Cisplatin 75mg/m2 IV over 60-120 minutes
  Other Names: No brands available
Drug: Bevacizumab — 5. Bevacizumab 15mg/kg IV over 90 minutes
  Other Names: Avastin

SUMMARY:
In the past, patients with advanced lung cancer who were inoperable underwent chemotherapy with one or more chemotherapeutic agents. More recently, novel new agents targeting specific enzymes or pathways responsible for cell division have been developed and clinicians have begun to utilize various combinations of these drugs with standard chemotherapeutic agents for the treatment of NSCLC. Some of these approaches have demonstrated a small but significant increase in survival among patients with advanced disease. Because a recently completed Phase 3 study of bevacizumab + Taxol/Carboplatin in first line NSCLC therapy demonstrated a 23% improvement in median survival, it would be appealing to see if a regimen of bevacizumab/ cisplatin/Alimta would also demonstrate a similar, or perhaps better, response rate.

DETAILED DESCRIPTION:
The majority of patients with NSCLC present with inoperable locally advanced or metastatic disease for which no curative therapy is available. For these patients, platinum based doublet combination regimens have become standard of care due to increased survival rates over platinum therapy alone.

In order to try to improve on the overall survival, clinicians have attempted to add a third cytotoxic agent to their standard regimen(s). Although this approach demonstrated an improved objective response, no additional benefit was noted in overall survival.

Recent development and approval of new targeted chemotherapies during the past 10 years has prompted clinical trials to test the efficacy of newly FDA approved agents such as gefitinib, erlotinib, and bevacizumab in advanced NSCLC.

Although gefitinib and erlotinib have both demonstrated clinical activity in refractory NSCLC, neither agent improved clinical outcome when added to standard 1st line platinum based chemotherapy. In contrast, a recently completed randomized Phase 3 trial investigating the addition of bevacizumab to 1st line paclitaxel plus carboplatin chemotherapy reported a 23% improvement in the median overall survival for the paclitaxel/carboplatin plus bevacizumab treatment arm (12.5m vs. 10.2m; p=0.007). It is therefore appealing to study a cisplatin combination with bevacizumab to determine if there is any additive benefit. Pemetrexed is an ideal agent to use in combination with cisplatin since it is well tolerated and efficacy is comparable to other cisplatin combinations. Patients will receive a maximum of 6 cycles. Those who complete 1 cycle will be evaluated for toxicity; more than 1 cycle, response.

ELIGIBILITY:
Inclusion Criteria:

* Have stage IIIB (malignant pleural or pericardial effusion) or stage IV disease.
* Be chemotherapy naïve.
* Have measurable disease by RECIST, defined as at least 1 lesion that can be accurately measured in at least 1 dimension as >20 mm with conventional techniques or >10 mm with spiral CT scan; the longest diameter is to be recorded.
* Are 18 years of age or older.
* Have a life expectancy greater than 3 months.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Are able to provide written informed consent in accordance with all applicable regulations and follow the study procedures. Patients must be capable of understanding the investigational nature, potential risks and benefits of the study.
* The ability to interrupt NSAIDS 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of Alimta and the ability to take folic acid, Vitamin B12 and dexamethasone according to protocol.

Exclusion Criteria:

* Have had prior chemotherapy (or an epidermal growth factor receptor (EGFR TKI) for treatment of advanced disease
* Intrathoracic lung carcinoma of squamous cell histology
* History of hemoptysis (bright red blood of 1/2 teaspoon or more per episode) within 1 month prior to study enrollment.
* Current, ongoing treatment with full-dose warfarin or its equivalent (i.e., unfractionated and/or low molecular weight heparin).
* Current or recent (within 10 days of enrollment) use of aspirin (>325 mg/day) or chronic use of other NSAIDs.
* Cardiovascular concerns.
* Have had radiation therapy within 2 weeks prior to enrollment.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1.
* Serious, non-healing wound, ulcer, or bone fracture.
* Have inadequate organ function at the Screening visit.
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation).
* Have uncontrolled active systemic infection requiring treatment.
* Have had treatment for a cancer other than NSCLC within 5 years prior to enrollment, with the exception of basal cell carcinoma or cervical cancer in situ.
* Have known human immunodeficiency virus (HIV) positive or hepatitis B surface antigen-positive status or known active hepatitis C infection. Patients assessed by the investigator to be at risk for HIV, hepatitis B or C infection should be tested in accordance with local regulations.
* Are a pregnant or breast-feeding female. Confirmation that the patient is not pregnant must be established by a negative serum Beta-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during the Screening Period. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Are unwilling to employ adequate means of contraception (condoms, diaphragm, birth control pills, injections, intrauterine device, or abstinence).
* Are currently receiving or have previously received an investigational agent for any reason within 4 weeks of enrollment.
* Presence of third space fluid which cannot be controlled by drainage.
* Inability to comply with study and/or follow-up procedures.
* Prior history of hypertensive crisis or hypertensive encephalopathy.
* History of stroke or transient ischemic attack within 6 months prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stoopler, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - North Shore University Hospital, Lake Success, New York
  - Columbia University Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twelve participants enrolled (signed a consent form). Two participants were screen failures and data was not collected for an additional two participants as the study terminated early, resulting in 8 participants starting the study.
Period: Overall Study
Arm/Group | Pemetrexed, Cisplatin, Bevacizumab
Started | 8
Completed | 0
Not Completed | 8
Not completed — Early Study Termination | 8

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed, Cisplatin, Bevacizumab
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Progression Free Survival (PFS)
Description: PFS defined as the time from the date of the first dose to the first date of disease progression or death.
Time Frame: Up to 1 year
Population: Data was NOT collected due to early study termination and therefore not analyzed.
Arm/Group | Pemetrexed, Cisplatin, Bevacizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Pemetrexed, Cisplatin, Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed, Cisplatin, Bevacizumab (N=8)
Elevated Creatinine (General disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Back Pain (General disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Chest Pain (General disorders) | 1
Pain (General disorders) | 1
Headache (General disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 4
Flank Pain (General disorders) | 1
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 1
Abdominal Pain (General disorders) | 2
Allergic Reaction (Immune system disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Pruritis (General disorders) | 1
Hypertension (Cardiac disorders) | 4
Hoarseness (General disorders) | 1
Anorexia (Gastrointestinal disorders) | 2
Epistaxis (General disorders) | 2
Anxiety (Psychiatric disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2
Hypocalcemia (Blood and lymphatic system disorders) | 1
Sore throat (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Epigastric Discomfort (Gastrointestinal disorders) | 1
Cough (General disorders) | 1
Hypokalemia (Blood and lymphatic system disorders) | 1
Increased Blood Urea Nitrogen (Blood and lymphatic system disorders) | 1
Urinary Tract Infection (Renal and urinary disorders) | 1
Left calf cramps (Musculoskeletal and connective tissue disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Vasovagal Reaction (General disorders) | 1
Taste Alteration (General disorders) | 1
Hyponatremia (Blood and lymphatic system disorders) | 1
Hypomagnesemia (Blood and lymphatic system disorders) | 1
Hypoglycemia (Blood and lymphatic system disorders) | 1
Periorbital edema (Eye disorders) | 1
Increased Nasal Mucus (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Runny Nose (General disorders) | 1
Conjunctivitis (Eye disorders) | 1
Skin Tears (Skin and subcutaneous tissue disorders) | 1
Weight Loss (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No